CLINICAL TRIAL: NCT02458833
Title: Home Plate: A Randomized Controlled Trial of a Community-Engaged Intervention to Improve Home Food Preparation Practices and Health During Early Childhood
Brief Title: Home Plate: A Trial to Improve Home Food Preparation Practices Among Parents of Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-011720
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: Obesity; Nutrition; Home Food Preparation; Home Food Environment; Peer Mentoring; Early Head Start; Cooking; Diet
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Behavioral: Home Plate intervention
  Interventions: Behavioral: Home Plate
- Delayed Entry Control (Experimental): This Arm will receive the Home Plate intervention 3 months after the Intervention Arm completes the intervention.
  Interventions: Behavioral: Home Plate

INTERVENTIONS:
Behavioral: Home Plate — Home Plate is a community-based, peer mentored intervention aimed at improving home food preparation practices in families with young children. Through 6 classes, this intervention explores topics related to regularly preparing healthy foods at home.

SUMMARY:
This study aims to test the effectiveness of a community-based, peer-mentored intervention to improve home food preparation practices in families with young children.

DETAILED DESCRIPTION:
Barriers to healthy eating and active living are at the heart of the obesity epidemic. This study focuses on a key factor underlying healthy eating: home food preparation. This study aims to test the effectiveness of a community-based, peer-mentored intervention to improve home food preparation practices in families with young children. The investigators will partner with community-based organizations serving families with children ages 1 to 3 years in West Philadelphia aiming specifically to:

1. Test the intervention's effect on diet and physical health.

   Hypothesis 1: The intervention group will have improved home food preparation practices and a healthier diet compared to the control group.
2. Test the intervention's effect on family health.

   Hypothesis 2: The intervention group will report improved parenting skills and more hopeful patterns of thinking.
3. Identify factors present at baseline and during engagement with the intervention that distinguish intervention participants who have improved diet, physical health, and family health from those who do not.

ELIGIBILITY:
Inclusion Criteria: mentees

1. English-speaking
2. Able to give informed consent.
3. Legal guardian and caregiver of at least one child, age 1-3 years

Inclusion Criteria: children

1. 1-3 year old children of mentee primary caregivers enrolled in the study
2. If a mentee caregiver has more than one child, then all their eligible children (ages 1-3 years) will be enrolled in the study.

Inclusion Criteria: peer mentors

1. Eligible peer mentors should meet the inclusion criteria set forth above for mentees. (Children of peer mentors will not be eligible for this study.)

   In addition,
2. The study team will decide which participants will be invited to be peer mentors, based on attributes including interest, leadership ability, and home food preparation skills.

Exclusion Criteria

1. Caregivers and children not meeting the inclusion criteria above.
2. Caregivers who are pregnant at the time of enrollment.
3. Caregivers or children with a medical condition that significantly affects their diet or eating habits. (The study team will ask during the time of recruitment if subjects or their children have a medical condition that significantly affects diet or eating habits.)
4. Subjects who, in the opinion of the Investigator, may be unable to participate in the study schedules or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-06; Primary Completion 2017-07 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
Dietary Energy Density (Child Participants) | 19-30 weeks from baseline
  Child participants' 24-hour dietary recalls will be collected by trained study staff from adult caregivers. 24-hour dietary recalls will be collected on a minimum of 2 and a maximum of 3 separate days. The results will then be used to calculate the energy density of the child's diet.

SECONDARY OUTCOMES:
Home Food Preparation Practices | 19-30 weeks from baseline
  Adult participants will complete surveys to assess the foods they usually prepare at home, as well as the time, energy, and confidence they have to prepare meals for their household.
Home Food Environment | 19-30 weeks from baseline
  Adult participants will complete surveys to assess the foods currently available in their homes, how they feel about managing food-related tasks, and the interactions they have with their child(ren) regarding food and eating.
Household Routines | 19-30 weeks from baseline
  Adult participants will complete surveys to assess their household routines related to activities such as sleep, physical activity, and screen time.
Emotional and Family Health | 19-30 weeks from baseline
  Adult participants will complete surveys to assess the their emotional health and the health of their families.
Body mass index | 19-30 weeks from baseline
  Heights and weights will be measured by trained study staff and will be used to calculate body mass index (BMI) of adult and child participants.
Dietary Energy Density (Adult Participants) | 19-30 weeks from baseline
  24-hour dietary recalls will be collected by trained study staff from adult study participants. 24-hour dietary recalls will be collected on a minimum of 2 and a maximum of 3 separate days. The results will then be used to calculate dietary energy density.
Diet Quality | 19-30 weeks from baseline
  In addition to dietary energy density, 24-hour dietary recall data will be used to calculate both child and adult study participants' intake of fruits, vegetables, whole grains, and added sugars.

CONTACTS AND LOCATIONS:
Overall Officials: Senbagam Virudachalam, MD, MSHP, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States